CLINICAL TRIAL: NCT02184806
Title: Autograft of Human Ovarian Tissue: Efficiency and Safety Evaluation
Brief Title: Autograft of Human Ovarian Tissue : Efficiency and Safety
Acronym: CAROLéLISA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P080802
Record Dates: First submitted 2014-06-13; First posted 2014-07-09 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Ovarian Tissue Transplantation
Keywords: Ovarian tissue transplantation; Cryopreserved ovarian tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1- orthotopic graft (Experimental)
  Interventions: Procedure: orthotopic graft
- 2- heterotopic graft (Experimental)
  Interventions: Procedure: heterotopic graft

INTERVENTIONS:
Procedure: orthotopic graft — (1) laparoscopy (2) ovarian fragments can be put back inside the pelvic cavity close to the natural location of the ovaries or
  Other Names: ovarian tissue autotransplantation
  Arms: 1- orthotopic graft
Procedure: heterotopic graft — 1. put under the skin
  2. the ovarian fragments can be put under the skin of the abdomen
  Arms: 2- heterotopic graft

SUMMARY:
Ovarian tissue cryopreservation is a new technique for female fertility preservation. One way to restore fertility is autotransplantation of ovarian tissue.

The principal purpose of this study will be to evaluate the efficiency and safety of this procedure.

DETAILED DESCRIPTION:
Ovarian tissue cryopreservation is a new technique for female fertility preservation before gonadotoxic treatments. The first ovarian tissue cryopreservations were performed 10 years ago. There are two main methods to use frozen ovarian cortex: autograft of ovarian fragments and in vitro follicular growth. At the present time, none mature oocytes were obtained after culture. Since 2000, around twenty publications stating autografts of ovarian cortex reported 8 pregnancy and 6 life birth of healthy babies.

Since 1998 until 2008, in the unit of reproduction biology of pitie-salpetriere hospital in Paris, France, 330 patients have had an ovarian tissue cryopreservation for fertility preservation before gonadotoxic treatment. Among them, at the present time, 180 have a procreative age and in consequence, could ask for the use of their ovarian cortex.

The general aim of this protocol will be to propose to women wishing to have a baby, an ovarian tissue transplantation if the patients have an premature ovarian failure.

The principal aim of this study will be to evaluate the efficiency and the safety of ovarian transplantation.

Before grafting, the absence of contra- indication will be check. An informed consent will be signed by the patient. Autograft of ovarian cortex will be performed either in orthotopic or in heterotopic localization according to the pathology and a possible contra-indication to orthotopic position.

After graft, each month hormonal assessment, ovarian echography and, after 3 months, an MRI, will be performed.

Assisted Reproductive Technologies (ART) will be performed in case of heterotopic graft and if necessary in case of orthotopic graft.

The efficiency of ovarian tissue autograft will be appreciated by the delay before the recovery of the ovarian function, the oocyte and embryos qualities in case of ART.

Finally, the number of pregnancies and live births will be also appreciated as well as a possible recurrence of the pathology.

ELIGIBILITY:
Inclusion criteria :

* adult women (age ≥ 18 years old) who stored ovarian fragments before gonadotoxic treatments
* Women who desire to conceive
* Married women or in stable couple
* Cured women or in remission
* Women suffering of Premature ovarian failure
* Consenting women
* women with health insurance

Exclusion criteria :

* age < 18 years
* women with normal ovarian function
* women with a disease at high risk for ovarian metastasis
* women with contraindication for surgery
* women with contraindication for pregnancy
* not cured women or not in remission
* women without health insurance

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Biological (FSH, LH, E2 and AMH) changes from graft until the revovery of ovarian function | every month after graft, up to 18 months
  FSH, LH, E2 and AMH follow up every month after graft until the recovery of ovarian function, up to 18 months
Radiological (ultrasonography and MRI) changes in ovarian imaging from graft until the revovery of ovarian function | every month after graft, up to 18 months
  Radiological (only ultrasonography the first 3 months and after ultrasonography and MRI) follow up every month after graft until the recovery of ovarian function, up to 18 months

SECONDARY OUTCOMES:
Graft vascularization | every month up to 18 months
Relapse of the pathology | every month up to 18 months
Delay and quality of the ovarian function recovery between ortho and heterotopic graft | after ovarian function recovery, up to 18 months
Number of ovarian fragments necessary for ovarian function recovery | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Poirot Catherine, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Tenon, service de Biologie de la reproduction, Paris, France

REFERENCES:
- [Derived] Vatel M, Torre A, Paillusson B, Scheffler F, Bergere M, Benkhalifa M, Le Martelot MT, Leperlier F, Mirallie S, Selleret L, Prades-Borio M, Neuraz A, Barraud-Lange V, Boissel N, Fortin A, Poirot C. Efficacy of assisted reproductive technology after ovarian tissue transplantation in a cohort of 11 patients with or without associated infertility factors. J Assist Reprod Genet. 2021 Feb;38(2):503-511. doi: 10.1007/s10815-020-02033-9. Epub 2021 Jan 3. PMID 33389379
- [Derived] Poirot C, Fortin A, Lacorte JM, Akakpo JP, Genestie C, Vernant JP, Brice P, Morice P, Leblanc T, Gabarre J, Delmer A, Badachi Y, Drouineaud V, Gouy S, Chalas C, Egels S, Dhedin N, Touraine P, Dommergues M, Lebegue G, Wolf JP, Capron F, Lefebvre G, Boissel N; CAROLeLISA Cooperative Group. Impact of cancer chemotherapy before ovarian cortex cryopreservation on ovarian tissue transplantation. Hum Reprod. 2019 Jun 4;34(6):1083-1094. doi: 10.1093/humrep/dez047. PMID 31116405